CLINICAL TRIAL: NCT07361432
Title: Improving Pain and Functioning Using an Integrative Digital Treatment for Chronic Pain and Addiction in Veterans With Opioid Use Disorder Receiving Buprenorphine
Brief Title: Digital Treatment for Chronic Pain and Addiction in Veterans With Opioid Use Disorder Receiving Buprenorphine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRDA-001-25M; 1I01RD000376-01A1 (Other Grant/Funding Number: ORD)
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Chronic Pain
Keywords: Buprenorphine; Chronic pain; Opioid-related disorders; Internet-based intervention; Cognitive behavioral therapy
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The present study is a hybrid type 1 effectiveness-implementation trial of IMPACT versus ETAU to improve functioning and quality of life in Veterans with chronic pain and OUD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMPACT (Experimental): Data from Veteran participants randomized to digital intervention (IMPACT)
  Interventions: Behavioral: Integrating the Management of Pain and Addiction via Collaborative Treatment (IMPACT)
- ETAU (Placebo Comparator): Data from Veteran participants randomized to ETAU (no access to IMPACT)
  Interventions: Behavioral: Enhanced Treatment as Usual (ETAU)

INTERVENTIONS:
Behavioral: Integrating the Management of Pain and Addiction via Collaborative Treatment (IMPACT) — The IMPACT program is a 9-module web-based treatment augmented with personalized weekly feedback from an expert coach for people with chronic pain and OUD receiving MOUD.
  Arms: IMPACT
Behavioral: Enhanced Treatment as Usual (ETAU) — ETAU is inclusive of medication management, groups, and individual treatment offered within the outpatient buprenorphine clinics at the study sites. Additionally, study staff will provide a a comprehensive list of pain, addiction and mental health treatment options that are specific to their VA facility.
  Arms: ETAU

SUMMARY:
Chronic pain is common in individuals with opioid use disorder (OUD) and the first-line treatment, Medication for OUD (MOUD), does not address the considerable functional impairments associated with chronic pain. Veterans with OUD and chronic pain could benefit from integrated, behavioral treatment for chronic pain and addiction, but VHA MOUD clinics often lack the resources to offer these services. The proposed study will examine the effectiveness of an evidence-based digital chronic pain and addiction treatment that Veterans can do from home, which can provide a flexible option for Veterans to engage in treatment from home and the Veterans Health Administration (VHA) a means to provide care without placing trained clinicians at each facility.

DETAILED DESCRIPTION:
The Integrating the Management of Pain and Addiction via Collaborative Treatment (IMPACT) is a 9-week, web-based treatment supplemented with daily digital surveys that inform personalized weekly feedback messages for people with chronic pain and OUD receiving MOUD. IMPACT is an integration of two previously tested technology-based interventions developed in a prior NIH-funded trial. Typically, VHA pain treatment resources are greater than civilian healthcare settings; therefore, the comparator group (enhanced treatment as usual or ETAU) in the current trial is a necessary step to rigorously test IMPACT specifically within Veteran Health Administration (VHA) clinical care.

ELIGIBILITY:
Inclusion Criteria:

* an ICD-11 OUD diagnosis in the VHA electronic health record (EHR)
* receipt of buprenorphine from outpatient addiction clinic with stable (i.e., unchanged in 2 weeks or since last injection) dose confirmed by the prescribing clinician. Both oral and injectable buprenorphine formulations will be eligible with dose stabilization required to isolate chronic pain from withdrawal-related pain associated with non-therapeutic dose
* presence of musculoskeletal pain that is bothersome or high-impact per the Graded Pain Scale - Revised
* access to a web-connected device to complete daily surveys and connect to IMPACT treatment site
* ability to participate safely in the walking portion of the intervention as evidenced by patient-reported ability to walk at least one block

Exclusion Criteria:

* dementia-related EHR diagnosis
* participant-reported vision or hearing impairments that would preclude use of the IMPACT system
* legal actions that would make study completion unlikely
* current or past 12 month engagement in CBT for chronic pain treatment
* planned surgical intervention for pain
* physical or mental health conditions that would interfere with ability to meaningful engage in IMPACT and MOUD treatment (e.g., uncontrolled bipolar disorder, active suicidal ideation, receipt of hospice or end-of-life palliative care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-11-02 (Estimated); Primary Completion 2029-06-03 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pain Interference 6b | 3-months post-randomization
  T-score will be calculated from raw scores with a mean of 50 and standard deviation of 10 (lower corresponds to less pain interference).

SECONDARY OUTCOMES:
PROMIS Pain Interference 6b | 6- and 9-months post randomization
  T-score will be calculated from raw scores with a mean of 50 and standard deviation of 10 (lower score corresponds to less pain interference).
Veterans Rand 12-Item Health Survey (VR-12) | 3-months post-randomization
  T-score will be calculated from raw scores with a mean of 50 and standard deviation of 10 (lower corresponds to better quality of life).
Activity Measure for Post-Acute Care (AM-PAC) | 3-months post-randomization
  Measure has two scales: Basic Mobility (range: 0-24) and Daily Activity (range: 0-24); on both scales higher scores corresponds to better performance.
PROMIS Sleep Disturbance 6a and Duration | 3-months post randomization
  T-score will be calculated from raw scores with a mean of 50 and standard deviation of 10 (lower score corresponds to less sleep disturbance).
Buprenorphine retention | 3-months post randomization
  retention is defined as both continuous and verified enrollment in MOUD in the 30 days prior to the specified timepoint. Continuous will be defined as having a continuously active buprenorphine prescription with a record of dispensing that includes the prior 30 days verified by Electronic Health Record. Retention will be a binary outcome with 1 = retained (conditions met) and 0 = not retained
Buprenorphine adherence | 3-months post randomization
  Timeline Follow-back will collect days of use for buprenorphine since last time point. During treatment period, weekly Timeline Follow-back adherence to buprenorphine will be compared to daily surveys and active buprenorphine prescription will be verified in Electronic Health Record (EHR). If a participant does not complete Timeline Follow-Back and/or has missing data in daily surveys or did not pick up buprenorphine as prescribed in EHR, the week will be considered non-adherent. Injectable buprenorphine will be verified in EHR and, if participant received injection as scheduled, they will be considered adherent. Mean adherent weeks will be calculated in each group; higher number corresponds to greater adherence.
Non-prescribed opiate use | 3-months post randomization
  Timeline Follow-back will collect days of non-prescribed opiate use since last time point. Weekly Timeline Follow-back non-prescribed opiate use will be collected during treatment period. Mean days of non-prescribed opiate use in a week will be calculated in each group; higher number corresponds to greater non-prescribed opiate use.

CONTACTS AND LOCATIONS:
Overall Officials: R. Ross MacLean, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (4):
- United States (4):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF